CLINICAL TRIAL: NCT06552754
Title: Cybersickness Prevention and Mitigation in Virtual Reality for Healthy Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10001975; 001975-HG
Record Dates: First submitted 2024-08-09; First posted 2024-08-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01-06

CONDITIONS: Healthy Volunteers; Virtual Reality
Keywords: Healthy Volunteers; Virtual Reality; cybersickness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention: Motion Reset (Experimental): Participate in virtual reality activities
  Interventions: Behavioral: Motion Reset
- No intervention (No Intervention)
- Placebo experience (Placebo Comparator): Participate in virtual reality activities
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Motion Reset — virtual reality-based experiential, sensory intervention
  Arms: Intervention: Motion Reset
Behavioral: Placebo — virtual reality-based experiential, sensory experience without intervention
  Arms: Placebo experience

SUMMARY:
Background:

People use virtual reality (VR) technology to play games, socialize, work, or receive medical care. Some people have "cybersickness" after using VR. Cybersickness is similar to motion sickness. Symptoms include eye strain, nausea, dizziness, or headache. The symptoms are usually mild and go away after the person stops using VR. New software called Motion Reset is being designed to reduce symptoms of cybersickness during VR use.

Objective:

To see if Motion Reset software can reduce cybersickness in people using VR.

Eligibility:

Healthy adults aged 18 to 60 years.

Design:

Participants will have 1 clinic visit that will last about 1 hour. They will answer questions about how they are feeling. They will learn how to use the VR headset and the handheld game controllers.

The study will be broken into 2 parts. For the first part, participants will be assigned to 1 of 3 groups:

Group 1 will participate in a VR experience designed to prevent cybersickness. They will view screens and move around while they press buttons on a controller.

Group 2 will participate in a VR experience that is not designed to prevent cybersickness. They will view screens and move around while they press buttons on a controller.

Group 3 will have no VR experience.

Participants will complete 2 questionnaires about their experiences in the first part of the study.

For the second part, all participants will spend up to 20 minutes playing a commercial VR game called Jurassic World Aftermath. Every few minutes, they will be asked if they are experiencing discomfort.

After playing the game, participants will complete 12 questionnaires about their experience....

DETAILED DESCRIPTION:
Study Description:

This study involves investigation of a virtual reality (VR) experience intended to prevent cybersickness (similar to motion sickness and eye strain) from use of virtual reality equipment. Participants will be randomly assigned to one of three arms: active intervention, placebo (a similar VR experience that does not engage sensory systems purported to underlie efficacy), or a notreatment control. Following the intervention, participants will play a VRbased game used in previous research to slowly induce moderate levels of cybersickness in some individuals. During play, we will assess self-reported feelings of discomfort. Participants will be allowed to stop playing at any time or will be asked to stop playing if discomfort reaches a certain threshold. Self-report data will be collected prior to and following the intervention.

Objectives:

Primary Objective: Evaluate efficacy of an approach for prevention of cybersickness symptoms when using virtual reality.

Secondary Objectives: Investigate individual difference factors associated with efficacy; assess mechanisms involved in treatment efficacy

Endpoints:

Primary Endpoint: Self-reported cybersickness symptoms on the Simulator Sickness Questionnaire

Secondary Endpoints: Self-reported cybersickness and duration of stimulus game play. Investigate individual difference factors associated with efficacy; assess mechanisms involved in treatment efficacy

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged 18-60
* Ability to read, speak, and write in English
* Normal or corrected-to-normal hearing
* Normal vision or corrected-to-normal without use of glasses. Contact lenses for corrective purposes are acceptable.

Ability to read, speak and write in English is a requirement because the VR-based study materials and assessment are only available in English and several of the key questionnaires for the study are not validated in other languages.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Reporting motion sickness propensity of 0, 9 or 10 on a 0-10 scale where 0 =never experience motion sickness and 10 = experience motion sickness very frequently (self-assessed by participants).
* Reporting a history of photo-sensitive seizure disorders, vestibular disorders and/or other conditions that may make participants prone to nausea, dizziness, vertigo, ataxia, or incoordination.
* Known pregnancy
* Reporting current use of medication or supplements that inhibit nausea, e.g., Zofran/ondansetron, Phenergan/promethazine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
self-reported cybersickness | during and after VR use
  Assessed on numerical scale

SECONDARY OUTCOMES:
discontinuation of VR use | during VR use
  decision to discontinue VR during active session

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - Iowa State University, Ames, Iowa
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001975-HG.html